CLINICAL TRIAL: NCT05198297
Title: The Hydrus® Microstent for Intraocular Pressure (IOP) Reduction in Mild to Moderate Open-Angle Glaucoma
Brief Title: Safety and Effectiveness of the Hydrus Microstent
Acronym: FRONTIER
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLI314-C002; CP 20-002 (Other: Ivantis)
Record Dates: First submitted 2022-01-03; First posted 2022-01-20 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Open Angle Glaucoma; Primary Open Angle Glaucoma; Pseudoexfoliation Glaucoma; Pigmentary Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle; Exfoliation Syndrome | interventions — Ophthalmologic Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Hydrus Microstent (Experimental): Hydrus Microstent implanted in the eye per the supplied Hydrus Microstent Instructions for Use and associated training. Only one eye (study eye) will be implanted.
  Interventions: Device: Hydrus Microstent; Procedure: Ophthalmic surgery

INTERVENTIONS:
Device: Hydrus Microstent — Minimally invasive glaucoma surgery device implanted into the Schlemm's canal of the eye to provide a natural outflow pathway for aqueous humor, leading to a reduction in intraocular pressure (IOP). The Hydrus Microstent is intended for lifetime use of the glaucoma patient.
Procedure: Ophthalmic surgery — Implantation of the Hydrus Microstent performed under either local or topical ophthalmic anesthesia

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of the Hydrus Microstent for lowering intraocular pressure (IOP) in pseudophakic patients with open-angle glaucoma for whom IOP is not sufficiently controlled on topical hypotensive medication and prior to incisional glaucoma surgery.

DETAILED DESCRIPTION:
Qualified subjects will undergo ocular hypotensive medication washout prior to implantation with the Hydrus Microstent. Following implantation on Day 0, subjects will attend 8 scheduled postoperative visits: Day 1, Week 1, Month 1, Month 3, Month 6, Month 12, Month 18, and Month 24.

A decision to terminate the study was made by the Sponsor arising from challenges with enrollment of the target study population, leading to suspension of enrollment and revision of the follow-up period to 12 months. The total duration of participation for each subject was approximately 13 months including the medication washout prior to implantation.

This study was initiated by Ivantis, Inc. Ivantis was acquired by Alcon Research, and Alcon assumed sponsorship of the study in November 2022.

ELIGIBILITY:
Inclusion Criteria:

* Early or moderate glaucomatous optic nerve damage;
* Uncomplicated cataract surgery with well centered posterior chamber IOL greater than or equal to 365 days prior to the screening visit;
* Inadequately controlled IOP;
* Shaffer angle grade III-IV in all four quadrants;
* Age appropriate minimum central endothelial cell density;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Diagnosis of acute angle closure, chronic angle closure, or congenital, malignant, or developmental glaucoma;
* Requires oral hypotensive medications;
* Shallow or flat anterior chamber;
* Prior glaucoma surgery;
* Ocular hypertension;
* Other protocol-defined exclusion criteria may apply.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Number of Subjects (Responders) with unmedicated DIOP greater than 6 mmHg and less than or equal to 21 mmHg with a reduction of greater than or equal to 20% from baseline and absence of secondary glaucoma surgery or loss of light perception | Baseline, Month 12 postoperative
  Intraocular pressure (IOP) will be measured using Goldmann tonometry. Three separate IOP measurements will be taken over an 8-hour period and averaged together to achieve mean diurnal intraocular pressure (DIOP). Baseline is defined as post ocular hypotensive medication washout and prior to Day 0, day of surgery. This is a co-primary endpoint. No hypothesis testing is prespecified.

SECONDARY OUTCOMES:
Mean Change in Unmedicated DIOP From Baseline to Month 12 and Absence of Secondary Glaucoma Surgery or Loss of Light Perception | Baseline, Month 12 postoperative
  IOP will be measured using Goldmann Applanation tonometry. Three separate IOP measurements will be taken over an 8-hour period and averaged together to achieve mean DIOP. Baseline will be defined as post ocular hypotensive medication washout and prior to Day 0, day of surgery. A negative change value represents an improvement. This is a co-primary endpoint. No hypothesis testing is prespecified.

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Clinical Project Lead, Surgical, Study Director — Alcon Research, LLC
Locations (5):
- United States (5):
  - Vold Vision PLLC, Bentonville, Arkansas
  - The Eye Clinic of Florida, Zephyrhills, Florida
  - Fraser Eye Care Center, Fraser, Michigan
  - Cincinnati Eye / Apex Eye, Mason, Ohio
  - Eye Centers Of Racine And Kenosha, Kenosha, Wisconsin

IPD SHARING:
Plan to Share IPD: No